CLINICAL TRIAL: NCT02924090
Title: Hyperventilation and ECT Seizure Duration: Effects on Cerebral Oxygen Saturation, and Therapeutic Outcome With Comparisons Between Etomidate and Ketamine in Patients With Major Depressive Disorder
Brief Title: Hyperventilation Combined With Etomidate or Ketamine Anesthesia in ECT Treatment of Major Depression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2015050
Record Dates: First submitted 2016-09-30; First posted 2016-10-05 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-09

CONDITIONS: Depression
Keywords: Major depressive disorder; Etomidate; Ketamine; Hyperventilation; Electroconvulsive therapy; Depression; Anesthesia; Nervous System Diseases; Mental Disorders; Electroencephalography; Cerebral Metabolism
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Hyperventilation; Nervous System Diseases; Mental Disorders | interventions — Etomidate; Ketamine; Electroconvulsive Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ECT with Etomidate (Active Comparator): Immediately prior to ECT study patients will be administered intravenous etomidate for anesthesia at a dose of 0.3 mg/kg given as a bolus dose.
  Interventions: Drug: Etomidate; Procedure: Electroconvulsive therapy (ECT)
- ECT with Ketamine (Active Comparator): Immediately prior to ECT study patients will be administered intravenous ketamine for anesthesia at a dose of 0.5 -1.0 mg/kg given as a bolus dose.
  Interventions: Drug: Ketamine; Procedure: Electroconvulsive therapy (ECT)
- ECT with Etomidate and Hyperventilation (Active Comparator): Immediately prior to ECT study patients will be administered intravenous etomidate for anesthesia at a dose of 0.3 mg/kg given as a bolus dose. Hyperventilation will be administered (20 breaths in 30 seconds) by face mask immediately prior to ECT.
  Interventions: Drug: Etomidate; Procedure: Hyperventilation; Procedure: Electroconvulsive therapy (ECT)
- ECT with Ketamine and Hyperventilation (Active Comparator): Immediately prior to ECT study patients will be administered intravenous ketamine for anesthesia at a dose of 0.5 -1.0 mg/kg given as a bolus dose. Hyperventilation will be administered (20 breaths in 30 seconds) by face mask immediately prior to ECT.
  Interventions: Drug: Ketamine; Procedure: Hyperventilation; Procedure: Electroconvulsive therapy (ECT)

INTERVENTIONS:
Drug: Etomidate — Etomidate will be administered as a bolus intravenously to induce an adequate depth of anesthesia just prior to ECT at a dose of 0.3 mg/kg
  Other Names: Amidate
  Arms: ECT with Etomidate; ECT with Etomidate and Hyperventilation
Drug: Ketamine — Ketamine will be administered as a bolus intravenously to induce an adequate depth of anesthesia just prior to ECT at a dose of 0.5 to 1.0 mg/kg.
  Other Names: Ketalar
  Arms: ECT with Ketamine; ECT with Ketamine and Hyperventilation
Procedure: Hyperventilation — Hyperventilation will be performed in patients after full pre-oxygenation and induction of anesthesia, by administering 20 breaths in 30 seconds using a well-fitting face mask immediately before application of the ECT electrical stimulus.
  Arms: ECT with Etomidate and Hyperventilation; ECT with Ketamine and Hyperventilation
Procedure: Electroconvulsive therapy (ECT) — Bilateral, bitemporal electrode placement will be utilized to elicit a seizure via a SpECTrun 5000Q (MECTA Inc.). The electrical dose required will be determined in advance by the patient's attending psychiatrist.

SUMMARY:
This is a randomized controlled study assessing the effect of pre-emptive hyperventilation on ECT seizure duration, cerebral desaturation and remission of depressive symptoms in patients with Major Depressive Disorder. Comparison of etomidate and ketamine on remission of depressive symptoms with and without pre-emptive hyperventilation will also be studied.

DETAILED DESCRIPTION:
Electroconvulsive therapy (ECT) is an effective treatment for medication-resistant forms of depression, including major depressive disorder and mania. Therapeutic success of ECT is related to the duration and quality of Electroencephalogram (EEG) and motor seizures. Previous studies have demonstrated that deliberate hyperventilation augments seizure duration in anesthetized subjects. It has also been shown that seizure activity significantly increases cerebral metabolic rate, predisposing the patient to potentially severe cerebral desaturation events. These desaturation events are predicted to be exacerbated by pre-emptive hyperventilation which has a potent cerebral vasoconstrictive effect. Despite the widespread use of ECT, little is known about the effect of hyperventilation on cerebral metabolism in this setting. Ketamine has recently been demonstrated to have anti-depressant properties in patients with major depressive disorder, suggesting that patients treated with ketamine anesthesia and then ECT, may benefit clinically from the additive effects of both treatment modalities, compared to ECT alone.

The investigators hypothesize that hyperventilation will facilitate prolonged seizure duration and faster remission of depressive symptoms. As well there may be significant cerebral desaturation and cardiovascular side effects of ECT therapy following hyperventilation. Lastly, the effect of hyperventilation on the efficacy of ECT therapy may be improved when ketamine anesthesia is used simultaneously. To test this hypothesis this study will compare ketamine anesthesia to etomidate anesthesia. Etomidate is a short acting anesthetic that is commonly used in these procedures.

The study objectives (primary and secondary) are as follows:

1. To quantify the effect of hyperventilation and type of anesthetic agent on ECT-induced seizure duration
2. To assess the effect of hyperventilation immediately prior to ECT on cerebral metabolism as measured by cerebral oximetry
3. To determine the effect of hyperventilation and anesthetic agent on the remission of symptoms in Major Depressive Disorder
4. To assess the side effect profile of hyperventilation during ECT on hemodynamics

ELIGIBILITY:
Inclusion Criteria:

* Adults patients aged 18 to 85 years
* Diagnosed with Major Depressive Disorder, unipolar or bipolar depression
* Undergoing ECT for treatment of their symptoms
* Currently residing in Manitoba

Exclusion Criteria:

* Relative contraindications to ECT therapy (recent MI or CVA, increased intracranial pressure, intracranial mass lesion, intracranial aneurysm, epilepsy, known cardiac arrhythmia, pheochromocytoma, pregnancy)
* Contraindications to etomidate (sepsis, primary or secondary adrenal insufficiency, porphyria)
* DSM-V diagnosis of a lifetime history of psychotic spectrum disorder
* Drug or alcohol dependence, or abuse within the past 3 months, soy-bean oil allergy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
EEG seizure duration (seconds) | Up to 3 minutes post ECT
  Duration of seizure spike wave morphology will be assessed by the attending psychiatrist and independently by a second psychiatrist.
ECT-induced seizure duration (seconds) | Up to 3 minutes post ECT
  Duration of motor seizures will be assessed by timing the onset and offset of appropriate motor twitches in the intrinsic foot muscles and extra-ocular muscles by the attending psychiatrist.

SECONDARY OUTCOMES:
Changes in cerebral metabolism assessed by cerebral saturation (%) | Up to 5 minutes post ECT
  Cerebral metabolism will be assessed by continuous cerebral oximetry measurements using the ForeSight Cerebral Oximeter, from immediately prior to ECT to 5 minutes post ECT
Remission of depressive symptoms assessed by HAM-D | Approximately one week prior to, and at 2, 4 and 8 weeks post ECT
  Patients will be assessed using a clinician-administered Hamilton Depression Rating Scale (HAM-D) both prior to, and at intervals of 2, 4 and 8 weeks after completion of the study. The HAM-D is a validated healthcare professional-administered assessments of clinical depressive symptoms including: hopelessness, guilt or depressed mood and physical symptoms such as agitation, restlessness and fatigue.
Remission of depressive symptoms assessed by MADRS | Approximately one week prior to, and at 2, 4 and 8 weeks post ECT
  Patients will be assessed using a clinician-administered Montgomery-Asberg Depression Scale (MADRS) both prior to, and at intervals of 2, 4 and 8 weeks after completion of the study. The MADRS is a validated healthcare professional-administered assessments of clinical depressive symptoms including: hopelessness, guilt or depressed mood and physical symptoms such as agitation, restlessness and fatigue.
Effect on blood pressure | Up to 7 minutes post ECT
  Systolic, diastolic and mean blood pressure will be recorded every minute from immediately prior to 7 minutes post ECT.
Effect on heart rate | Up to 7 minutes post ECT
  Heart rate (bpm) will be continuously recorded from immediately prior to 7 minutes post ECT.
Duration of stay in post-anesthesia care unit (hours) | Up to 2 hours post arrival in post-anesthesia care unit (PACU).
Incidence of nausea in post-anesthesia care unit (%) | Up to 2 hours post arrival in PACU.
  The number of instances of nausea while in PACU will be recorded.
Incidence of vomiting in post-anesthesia care unit (%) | Up to 2 hours post arrival in PACU.
  The number of instances of vomiting while in PACU will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ian McIntyre, MD, MSc, Principal Investigator — University of Manitoba; Michael Harrington, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loo C, Simpson B, MacPherson R. Augmentation strategies in electroconvulsive therapy. J ECT. 2010 Sep;26(3):202-7. doi: 10.1097/YCT.0b013e3181e48143. PMID 20562640
- [Background] Aksay SS, Bumb JM, Janke C, Hoyer C, Kranaster L, Sartorius A. New evidence for seizure quality improvement by hyperoxia and mild hypocapnia. J ECT. 2014 Dec;30(4):287-91. doi: 10.1097/YCT.0000000000000109. PMID 24625713
- [Background] Fabbri F, Henry ME, Renshaw PF, Nadgir S, Ehrenberg BL, Franceschini MA, Fantini S. Bilateral near-infrared monitoring of the cerebral concentration and oxygen-saturation of hemoglobin during right unilateral electro-convulsive therapy. Brain Res. 2003 Dec 5;992(2):193-204. doi: 10.1016/j.brainres.2003.08.034. PMID 14625058
- [Background] Ghasemi M, Kazemi MH, Yoosefi A, Ghasemi A, Paragomi P, Amini H, Afzali MH. Rapid antidepressant effects of repeated doses of ketamine compared with electroconvulsive therapy in hospitalized patients with major depressive disorder. Psychiatry Res. 2014 Feb 28;215(2):355-61. doi: 10.1016/j.psychres.2013.12.008. Epub 2013 Dec 13. PMID 24374115